CLINICAL TRIAL: NCT05756049
Title: Procalcitonin Protocol Use to Guide Antibiotic Therapy Duration in the Intensive Care Unit
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 117.PHA.2022.R
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Comparing Antibiotic Duration of Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: compare antibiotic duration of therapy — To compare antibiotic duration of therapy before and after the implementation of the PCT protocol in the ICU.

SUMMARY:
To compare and contrast antibiotic use and its effects on patient outcomes before and after the implementation of a PCT protocol in the ICU at Methodist Richardson Medical Center (MRMC).

DETAILED DESCRIPTION:
Based on previous clinical trials, current literature supports the use of PCT levels in combination with clinical assessments to help determine optimal antibiotic therapy. On May 30, 2022, MRMC launched a PCT protocol in the ICU that allows clinical pharmacy specialists to order PCT levels in certain bacterial infections. In order to determine the effects of the protocol, a retrospective quasi-experimental review will be conducted

ELIGIBILITY:
Inclusion Criteria:

* ● Patients aged 18 years or older

  * Patients being monitored on the PCT protocol
  * ICU location status for at least part of the admission
  * Received antibiotics in the ICU for a diagnosis of:

    * Community-acquired pneumonia
    * Hospital-acquired pneumonia
    * Ventilator-associated pneumonia
    * Sepsis and/or septic shock
    * Uncomplicated bacteremia with known source
    * Chronic obstructive pulmonary disorder exacerbation
    * Asthma exacerbation

Exclusion Criteria:

* Received antibiotics in the ICU for a diagnosis of:

  * Uncomplicated skin and soft tissue infections
  * Abscess
  * Empyema
  * Bacterial infections that require prolonged antibiotic therapy (e.g., osteomyelitis, endocarditis, tuberculosis, etc.)
  * Intra-abdominal infection
  * Urinary tract infection
  * Bacterial meningitis

    * Estimated Glomerular Filtration Rate <15 mL/min
    * Requiring renal replacement therapy
    * Status post cardiac arrest/target temperature management

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older Patients being monitored on the PCT protocol
  * ICU location status for at least part of the admission
  * Received antibiotics in the ICU for a diagnosis of:
    * Community-acquired pneumonia
    * Hospital-acquired pneumonia
    * Ventilator-associated pneumonia
    * Sepsis and/or septic shock
    * Uncomplicated bacteremia with known source
    * Chronic obstructive pulmonary disorder exacerbation
    * Asthma exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-11-29 (Estimated)

PRIMARY OUTCOMES:
Total days of antibiotic therapy | 6 months
  Actual antibiotic days and predicted antibiotic days (i.e., SAAR)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Richow, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Richardson Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All information will be blinded in compliance with GCP. The investigator will make all possible efforts to ensure compliance with all policies regarding sharing of PHI or research information. Only de-identified PHI will be shared in relevant research mediums. Data obtained from this research will be presented at the Texas Society of Health-System Pharmacists 2023 Alcalde Annual Seminar. The conference will be held on April 21st-23rd, 2023. Data obtained from this research will also be written in manuscript format and submitted to a peer-reviewed journal.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 1 year

REFERENCES:
- [Background] Magill SS, O'Leary E, Ray SM, Kainer MA, Evans C, Bamberg WM, Johnston H, Janelle SJ, Oyewumi T, Lynfield R, Rainbow J, Warnke L, Nadle J, Thompson DL, Sharmin S, Pierce R, Zhang AY, Ocampo V, Maloney M, Greissman S, Wilson LE, Dumyati G, Edwards JR, Chea N, Neuhauser MM; Emerging Infections Program Hospital Prevalence Survey Team. Assessment of the Appropriateness of Antimicrobial Use in US Hospitals. JAMA Netw Open. 2021 Mar 1;4(3):e212007. doi: 10.1001/jamanetworkopen.2021.2007. PMID 33734417
- [Background] Rice LB. Antimicrobial Stewardship and Antimicrobial Resistance. Med Clin North Am. 2018 Sep;102(5):805-818. doi: 10.1016/j.mcna.2018.04.004. Epub 2018 Jul 14. PMID 30126572
- [Background] Becker KL, Nylen ES, White JC, Muller B, Snider RH Jr. Clinical review 167: Procalcitonin and the calcitonin gene family of peptides in inflammation, infection, and sepsis: a journey from calcitonin back to its precursors. J Clin Endocrinol Metab. 2004 Apr;89(4):1512-25. doi: 10.1210/jc.2002-021444. No abstract available. PMID 15070906
- [Background] Schuetz P, Albrich W, Mueller B. Procalcitonin for diagnosis of infection and guide to antibiotic decisions: past, present and future. BMC Med. 2011 Sep 22;9:107. doi: 10.1186/1741-7015-9-107. PMID 21936959
- [Background] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Background] Schuetz P, Christ-Crain M, Thomann R, Falconnier C, Wolbers M, Widmer I, Neidert S, Fricker T, Blum C, Schild U, Regez K, Schoenenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Mueller B; ProHOSP Study Group. Effect of procalcitonin-based guidelines vs standard guidelines on antibiotic use in lower respiratory tract infections: the ProHOSP randomized controlled trial. JAMA. 2009 Sep 9;302(10):1059-66. doi: 10.1001/jama.2009.1297. PMID 19738090
- [Background] de Jong E, van Oers JA, Beishuizen A, Vos P, Vermeijden WJ, Haas LE, Loef BG, Dormans T, van Melsen GC, Kluiters YC, Kemperman H, van den Elsen MJ, Schouten JA, Streefkerk JO, Krabbe HG, Kieft H, Kluge GH, van Dam VC, van Pelt J, Bormans L, Otten MB, Reidinga AC, Endeman H, Twisk JW, van de Garde EMW, de Smet AMGA, Kesecioglu J, Girbes AR, Nijsten MW, de Lange DW. Efficacy and safety of procalcitonin guidance in reducing the duration of antibiotic treatment in critically ill patients: a randomised, controlled, open-label trial. Lancet Infect Dis. 2016 Jul;16(7):819-827. doi: 10.1016/S1473-3099(16)00053-0. Epub 2016 Mar 2. PMID 26947523
- [Result] Fridkin S, Baggs J, Fagan R, Magill S, Pollack LA, Malpiedi P, Slayton R, Khader K, Rubin MA, Jones M, Samore MH, Dumyati G, Dodds-Ashley E, Meek J, Yousey-Hindes K, Jernigan J, Shehab N, Herrera R, McDonald CL, Schneider A, Srinivasan A; Centers for Disease Control and Prevention (CDC). Vital signs: improving antibiotic use among hospitalized patients. MMWR Morb Mortal Wkly Rep. 2014 Mar 7;63(9):194-200. PMID 24598596